CLINICAL TRIAL: NCT01962012
Title: Effect of AcceleDent® Aura on Orthodontic Tooth Movement With Aligners
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoAccel Technologies Inc. (Industry)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OA-03
Record Dates: First submitted 2013-10-08; First posted 2013-10-14 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Malocclusion
Keywords: Orthodontic; Orthodontic Treatment; Accelerated Tooth Movement; Malocclusion; Device; AcceleDent Aura; Clear Aligners
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AcceleDent Aura (Experimental): AcceleDent Aura device provides a light vibration at 0.25 Newtons and 30 Hz frequency for 20 minutes daily.
  Interventions: Device: AcceleDent Aura
- Sham Device (Sham Comparator): Sham devices will look identical to active devices but will not deliver vibration to the patient.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: AcceleDent Aura
  Arms: AcceleDent Aura
Device: Sham Device
  Arms: Sham Device

SUMMARY:
The purpose of this study is to examine the amount of tooth movement achieved over time between subjects undergoing aligner treatment using a pulsation device known as AcceleDent® Aura with those not using the device.

DETAILED DESCRIPTION:
There are many variables that can affect the rate of tooth movement. Preliminary data showed that the rate of tooth movement may be affected by variables such as age, sex, as well as alveolar bone levels, tooth root length and alveolar bone quality. The purpose of this study is to examine the amount of tooth movement achieved over time between subjects undergoing aligner treatment using a pulsation device known as AcceleDent® Aura with those not using the device.

A preliminary validation pilot study will be done to calibrate all staff on study procedures. The pilot will consist of 3 subjects using the active AcceleDent® Aura device and 3 using the sham control AcceleDent® Aura device for 4 weeks. Study staff will be calibrated for all study procedures.

The primary study will be a prospective, single-center, randomized crossover clinical trial comparing two groups of subjects with 40 participants. Subjects will be randomized to groups that will receive aligner treatment while using either an active AcceleDent® Aura device or a sham control AcceleDent® Aura device for the first 6 weeks of the study. After 6 weeks, groups will cross-over and switch devices, and tooth movement will be followed for another 6 weeks. Patients will be blinded as to which device they are using. Amount of tooth movement per week, pain perception, and change in gingival crevicular fluid biomarkers will be outcomes assessed. Device safety evaluation to be performed will include adverse events and clinical examination findings including pulp vitality testing and periodontal probe results.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between and including the ages of 18 and 40 yo desiring orthodontic treatment that could be completed within two years of treatment with either fixed appliances or aligner treatment. Subjects may have had previous orthodontic procedures.
* Adult dentition with all upper front teeth present and any premolar and molar combination in the upper posterior of two teeth on each side.
* At least one upper maxillary central incisor that is positioned to allow anterio-posterior (AP) movement (crown tipping only) of 1.98 mm.
* Normal pulp vitality and healthy periodontal tissues as determined by intraoral exam.
* Good health as determined by medical history.
* Willingness and ability to comply with study procedures, attend study visits, and complete the study.
* The ability to understand and sign a written informed consent form, which must be signed prior to initiation of study procedures.

Exclusion Criteria:

* Severe malocclusions that would take longer than 2 years of treatment or require surgical intervention.
* Significant periodontal disease (> 3mm pocket depth or >1 mm of recession on upper anterior teeth).
* Active caries not under care of either a dentist or periodontist.
* Chronic daily use of any non-steroidal anti-inflammatory medication, estrogen, calcitonin, or corticosteroids.
* History of use or current use of any bisphosphonate medication or other medication for treatment of osteoporosis.
* Current smoker (must not have smoked in the last 6 months).
* Women may not be pregnant. Negative urine pregnancy tests prior to exposure to cone beam imaging is required to verify pregnancy status.
* Any condition or use of medication which in the opinion of the investigator interferes with the biology of tooth movement.
* Any condition which in the opinion of the investigator results in increased risk to the subject.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Rate of Orthodontic Tooth Movement (mm/week) | 12 Weeks

SECONDARY OUTCOMES:
Pain (Visual Analog Scale) | 3 Days After Receiving New Aligner

CONTACTS AND LOCATIONS:
Overall Officials: Timothy T Wheeler, DMD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Department of Orthodontics, Gainesville, Florida, United States